CLINICAL TRIAL: NCT07043998
Title: Evaluation of Full Veneered Porcelain-Fused-to-Metal Crowns Cemented With Self-Adhesive Resin Cement Using Two Curing Modes: A Randomized Clinical Trial
Brief Title: Evaluation of Full Veneered Porcelain-Fused-to-Metal Crowns Cemented With Self-Adhesive Resin Cement Using Two Curing Modes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Nabil, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24/5/25
Record Dates: First submitted 2025-06-11; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Restoration of Posterior Tooth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult patients requiring PFM crown cemented with dual cured self adhesive resin cement (Active Comparator)
  Interventions: Other: Self-adhesive resin cement in DUAL-CURED mode
- Adult patients requiring PFM crown cemented with self cured self adhesive resin cement (Active Comparator)
  Interventions: Other: Self-adhesive resin cement in SELF-CURED mode

INTERVENTIONS:
Other: Self-adhesive resin cement in SELF-CURED mode — PFM crowns veneered with porcelain system cemented using self-adhesive resin cement in SELF-CURED mode
  Arms: Adult patients requiring PFM crown cemented with self cured self adhesive resin cement
Other: Self-adhesive resin cement in DUAL-CURED mode — PFM crowns veneered with porcelain system cemented using self-adhesive resin cement in DUAL-CURED mode
  Arms: Adult patients requiring PFM crown cemented with dual cured self adhesive resin cement

SUMMARY:
P - Population/Patient Problem Adult patients requiring full coverage porcelain-fused-to-metal (PFM) crown restorations I - Intervention PFM crowns veneered with porcelain system cemented using self-adhesive resin cement in DUAL-CURED mode (light-cured for 20 seconds per surface) C - Comparison PFM crowns veneered with porcelain system cemented using self-adhesive resin cement in SELF-CURED mode (no light curing, 5 minutes self-cure) O - Outcome(s)

* Primary: Retention of PFM crowns (Modified USPHS criteria)
* Secondary: Marginal adaptation, recurrent caries, marginal discoloration (Modified USPHS criteria) T - Time 18-month follow-up period with evaluations at baseline, 6, 12, and 18 months

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients requiring full coverage PFM crown restorations
2. Age ≥ 21 years
3. Vital or endodontically treated teeth
4. Sufficient tooth structure for crown retention
5. Willing and able to provide written informed consent
6. Ability to attend all follow-up appointments
7. Adequate oral hygiene as determined by the investigator

Exclusion Criteria:

1. Patients with active periodontal disease (probing depth > 4mm, bleeding on probing)
2. Patients with severe parafunctional habits (e.g., bruxism confirmed by clinical examination)
3. Poor oral hygiene (plaque index > 30%)
4. Pregnancy or nursing
5. Systemic diseases affecting treatment outcomes (e.g., uncontrolled diabetes, immunosuppression)
6. Known allergies to study materials (metal alloys, porcelain, or resin cement components)
7. Inability to comply with study requirements
8. Current participation in other dental clinical trials
9. Active orthodontic treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Retention of PFM crowns | 18 months
  Modified USPHS criteria (Scores)

SECONDARY OUTCOMES:
Marginal adaptation | 18 months
  Modified USPHS criteria ( scores)
Recurrent caries | 18 months
  Modified USPHS criteria ( scores)
Marginal discoloration | 18 months
  Modified USPHS criteria ( scores)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No